CLINICAL TRIAL: NCT03492814
Title: Comparing the Effect of Different Suture Techniques on the Post Operative Morbidity After Surgical Removal of Impacted Mandibular Third Molar- A Randomized Clinical Study
Brief Title: Comparing Different Suturing Techniques on the Post-operative Morbidity After Removal of Impacted Mandibular Third Molar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melaka Manipal Medical College (Other)
Responsible Party: Principal Investigator, Abdul Kalam Azad, Assistant Professor, Dept Of Oral and Maxillofacial Surgery, Melaka Manipal Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MMMC/FOD/AR/B4/E C-2016(24)
Record Dates: First submitted 2018-04-01; First posted 2018-04-10 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Swelling; Trismus
Keywords: impacted third molar; suturing; post-operative morbidity
MeSH Terms: conditions — Trismus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partial wound closure (Experimental): 3 sutures distal to second molar and leaving the vertical releasing incision open without any sutures.
  Interventions: Procedure: partial wound closure
- Total wound closure (Active Comparator): 5 interrupted sutures with 2 sutures closing the vertical releasing incision and 3 sutures distal to second molar leading to a complete hermetic closure of the wound.
  Interventions: Procedure: total wound closure

INTERVENTIONS:
Procedure: partial wound closure — 3 sutures distal to second molar and leaving the vertical releasing incision open without any sutures.
  Arms: Partial wound closure
Procedure: total wound closure — 5 interrupted sutures with 2 sutures closing the vertical releasing incision and 3 sutures distal to second molar leading to a complete hermetic closure of the wound.
  Arms: Total wound closure

SUMMARY:
This study compares the effect of two types of suturing techniques in the postoperative swelling and mouth opening after surgical removal of impacted mandibular third molar. total wound closure will be performed in one group of participants while partial closure will be performed in the other group.

DETAILED DESCRIPTION:
Third molar surgeries are mostly associated with pain, swelling and limited mouth opening, referred to as post-operative morbidity. Wound closure technique is an operative factor which is associated with reduced post-operative morbidity. In the total wound closure, the mucoperiosteum is hermetically sealed whereas in the partial wound closure, a window or opening is left to allow for secondary healing. This study therefore compares the effect of partial and total wound closure techniques after surgical extraction of impacted mandibular third molar teeth in reducing the swelling and limited mouth opening.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing surgical removal of mesioangular impacted mandibular third molar.
* Healthy patients (ASA I) or patients with mild systemic disease with no functional limitations (ASA II).
* patients who are not allergic to the drugs and local anesthetic agent used in the surgical protocol.

Exclusion Criteria:

* Patients having systemic conditions that might have an effect on the bone growth or periodontal healing.
* patients who are on antibiotics premedication or any drugs that might affect wound healing.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03-10 (Actual); Primary Completion 2018-03-10 (Actual); Study Completion 2018-03-10 (Actual)

PRIMARY OUTCOMES:
change in the Measurement of mouth opening | baseline( preoperative) and 3rd and 7th day postoperatively.
  mouth opening is measure by measuring the maximum interincisal distance from the incisal edge of maxillary right central incisor to the incisal edge of the lower right central incisor using a vernier calliper in mm.
postoperative swelling | baseline ( preoperative) and 3rd and 7th day postoperatively.
  three line measurements were performed in cm using a measuring tape and mean was taken

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Kalam Azad, MDS, Principal Investigator — Melaka Manipal Medical College
Locations (1):
- Melaka Manipal Medical College, Malacca, Malaysia